CLINICAL TRIAL: NCT01098461
Title: A Dose Finding Study of GSK716155 Versus Placebo in the Treatment of Type 2 Diabetes Mellitus
Brief Title: Dose Ranging Study of Albiglutide in Japanese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110932
Record Dates: First submitted 2010-02-12; First posted 2010-04-02 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: dose-ranging; pharmacokinetics; GSK716155; Japan; albiglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- albiglutide 15mg weekly (Active Comparator): once weekly subcutaneous injection of albiglutide 15mg
  Interventions: Biological: albiglutide
- albiglutide 30mg weekly (Active Comparator): once weekly subcutaneous injection of albiglutide 30mg
  Interventions: Biological: albiglutide
- albiglutide 30mg every other week (Active Comparator): subcutaneous injection of 30mg albiglutide every other week
  Interventions: Biological: albiglutide
- placebo (Placebo Comparator): once weekly subcutaneous injection of placebo to match albiglutide
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: albiglutide — subcutaneous injection of albiglutide
  Other Names: placebo; albiglutide 30mg weekly; albiglutide 15mg weekly; albiglutide 30mg every other week
  Arms: albiglutide 15mg weekly; albiglutide 30mg every other week; albiglutide 30mg weekly
Biological: placebo — subcutaneous injection of placebo to match albiglutide
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, 4-parallel-group, dose ranging study evaluating the dose response, efficacy and safety of subcutaneously injected GSK716155 (albiglutide) in Japanese subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a Phase IIb, randomized, double-blind, placebo-controlled, multicenter, 4-parallel-group, dose ranging, superiority study evaluating the dose response, efficacy and safety of weekly and every other week subcutaneously injected GSK716155 (albiglutide) in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a historical diagnosis of type 2 diabetes mellitus who is currently treated with diet and exercise only or one OAD
* BMI ≥18 kg/m2 and <35 kg/m2 at Screening
* HbA1c between 7.0% and 10.0%, inclusive
* Fasting C-peptide ≥0.8 ng/mL (≥0.26 nmol/L)
* Female subjects of childbearing potential must be practicing adequate contraception .
* Able and willing to monitor his/her own blood glucose concentrations with a home glucose monitor.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* Uncorrected thyroid dysfunction
* Previous use of insulin within one month prior to screening, or more than seven total days of insulin treatment within three months prior to screening
* Clinically significantly cardiovascular and/or cerebrovascular disease including, but not limited to the following:

  * Previous history of stroke or transient ischemic attack
  * Active, unstable coronary heart disease within the past six months before Screening
  * Documented myocardial infarction within one year before Screening
  * Any cardiac surgery including percutaneous transluminal coronary angioplasty, coronary stent placement, or coronary artery bypass graft surgery within one year before Screening
  * Unstable angina
  * Clinically significant arrhythmia or valvular heart disease
  * Current heart failure NYHA class II to IV
  * Resting systolic pressure >160 mm Hg or diastolic pressure >95 mm Hg at Screening
  * ECG criteria at Screening
* Heart rate: <40 and >110 bpm
* PR interval: <120 and > 210 msec
* QRS interval: <70 and >120 msec
* QTc interval (Bazett): >450 msec or >480 msec with bundle branch block
* Fasting triglyceride level >400 mg/dL at Screening
* AST or ALT >2xULN, ALP and bilirubin >1.5xULN (except known Gilbert's syndrome and a fractionated bilirubin that shows conjugated bilirubin <35% of total bilirubin)
* If female, is currently lactating, within 6 weeks post-partum, pregnant, or actively trying to become pregnant
* Has significant renal disease as manifested by one or more of the following:

  * Creatinine clearance at screening <60 mL/min (calculated by Cockcroft-Gault formula) at Screening
  * Known loss of a kidney either by surgical ablation, injury or disease level
* A hemoglobinopathy that may affect determination of HbA1c level
* History of treated diabetic gastroparesis
* History of significant gastrointestinal surgery, including gastric bypass and banding, or surgeries thought to significantly affect upper gastrointestinal function
* Current ongoing symptomatic biliary disease or history of acute/chronic pancreatitis.
* Lipase and amylase at Screening > ULN
* Severe diabetic neuropathy, preproliferative retinopathy or proliferative retinopathy, history of ketoacidosis or hyperosmolar coma
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 3 years before Screening. (A history of treated cervical intraepithelial neoplasia I or cervical intraepithelial neoplasia II is allowed)
* Acute or chronic history of liver disease, positive hepatitis B surface antigen (HBsAg) or positive hepatitis C testing at Screening
* Current and history of alcohol or substance abuse
* Clinically significant anaemia or any other abnormal haematological profile that is considered by the investigator to be clinically significant
* Prior use of a GLP-1 analog
* Known allergy to any formulation excipients, or Baker's yeast, or history of drug, or other allergy which, in the opinion of the responsible study physician, contradicts participation
* History of or family history of medullary carcinoma of the thyroid.
* History of or family history of multiple endocrine neoplasia type 2
* Receipt of any investigational drug within the 12 weeks before Screening

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Japan (15):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- [Derived] Seino Y, Inagaki N, Miyahara H, Okuda I, Bush M, Ye J, Holland MC, Johnson S, Lewis E, Nakajima H. A randomized dose-finding study demonstrating the efficacy and tolerability of albiglutide in Japanese patients with type 2 diabetes mellitus. Curr Med Res Opin. 2014 Jun;30(6):1095-106. doi: 10.1185/03007995.2014.896327. Epub 2014 Mar 11. PMID 24552155
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria and completed a 4- to 8-week Run-in Period were then randomized to a 16-week Treatment Period, followed by an 8-week Follow-up Period. A total of 215 participants were randomized, and 212 received >=1 treatment dose.
Groups:
- Placebo: Participants received albiglutide-matching placebo administered via subcutaneous injection once a week via a fully disposable pen injector system for 16 weeks. The preferred post-rescue add-on treatment was insulin. Other medications may have been added at the investigator's discretion.
- Albiglutide 15 mg Weekly: Participants received albiglutide 15 milligrams (mg) administered via subcutaneous injection once a week via a fully disposable pen injector system for 16 weeks. The preferred post-rescue add-on treatment was insulin. Other medications may have been added at the investigator's discretion.
- Albiglutide 30 mg Weekly: Participants received albiglutide 30 mg administered via subcutaneous injection once a week via a fully disposable pen injector system for 16 weeks. The preferred post-rescue add-on treatment was insulin. Other medications may have been added at the investigator's discretion.
- Albiglutide 30 mg Every Other Week: Participants received albiglutide 30 mg or matching placebo administered via subcutaneous injection on alternating weeks via a fully disposable pen injector system for 16 weeks. The preferred post-rescue add-on treatment was insulin. Other medications may have been added at the investigator's discretion.
Period: Treatment Period (TP) (16 Weeks)
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Started | 53 | 52 | 54 | 53
Completed | 41 | 45 | 53 | 50
Not Completed | 12 | 7 | 1 | 3
Not completed — Persistent Hypoglycemia | 10 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Transferred to Oita (Japan) | 0 | 1 | 0 | 0
Period: Follow-up (FU) Period (8 Weeks)
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Started | 52 (Par. withdrawing from the TP could enter the FU Period. One par. did not participate in the FU.) | 52 | 53 (Par. withdrawing from the TP could enter the FU Period. One par. did not participate in the FU.) | 52 (Par. withdrawing from the TP could enter the FU Period. One par. did not participate in the FU.)
Completed | 52 | 49 | 52 | 52
Not Completed | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Transferred to Oita (Japan) | 0 | 1 | 0 | 0
Not completed — Follow-up Not Conducted Due to Earthquak | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week | Total
Number analyzed (Participants) | 53 | 52 | 54 | 53 | 212
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data are reported for members of the Safety Population, comprised of all enrolled participants who received at least one dose of study treatment. Participants were analyzed according to treatment received.
  Years | 57.5 (11.06) | 53.3 (10.29) | 58.0 (9.30) | 59.1 (8.49) | 57.0 (10.00)
Gender [Count of Participants; unit: Participants] — Baseline data are reported for members of the Safety Population, comprised of all enrolled participants who received at least one dose of study treatment. Participants were analyzed according to treatment received.
  Participants
    Female | 16 | 20 | 16 | 12 | 64
    Male | 37 | 32 | 38 | 41 | 148
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data are reported for members of the Safety Population, comprised of all enrolled participants who received at least one dose of study treatment. Participants were analyzed according to treatment received.
  participants
    Asian - Japanese Heritage | 53 | 52 | 54 | 53 | 212

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 16
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the value at Week 16 minus the value at Baseline. Based on Analysis of Covariance (ANCOVA): Change = treatment + Baseline HbA1c + prior therapy. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Week 16
Population: Intent-to-Treat (ITT) Population: all randomized participants with at least one post-Baseline assessment of the primary endpoint, HbA1c. Only those participants with a value available at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were discontinued from active treatment before Week 16.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Number analyzed (Participants) | 50 | 52 | 54 | 53
Percentage of HbA1c in the blood | 0.28 (0.099) | -0.61 (0.097) | -1.27 (0.095) | -0.82 (0.096)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 15 mg Weekly; Test type: Non-Inferiority or Equivalence — The p-value is from a two-sided t-test for the difference in means. Dunnett's method is used to adjust for multiple comparisons; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-1.22 to -0.57]
Statistical Analysis 2: Comparison: Placebo vs Albiglutide 30 mg Weekly; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-1.88 to -1.23]
Statistical Analysis 3: Comparison: Placebo vs Albiglutide 30 mg Every Other Week; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-1.43 to -0.78]

2. Secondary Outcome: Change From Baseline in HbA1c at Weeks 4, 8, 12, and 16
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the value at Week 16 minus the value at Baseline. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline; Week 4, Week 8, Week 12, and Week 16
Population: ITT Population with LOCF. Only those participants with a value available at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were discontinued from active treatment before Week 16.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Number analyzed (Participants) | 50 | 52 | 54 | 53
Percentage of HbA1c in the blood
  Week 4 | 0.03 (0.349) | -0.33 (0.301) | -0.61 (0.377) | -0.36 (0.383)
  Week 8 | 0.20 (0.628) | -0.59 (0.430) | -1.07 (0.578) | -0.74 (0.618)
  Week 12 | 0.24 (0.730) | -0.71 (0.464) | -1.26 (0.649) | -0.84 (0.720)
  Week 16 | 0.27 (0.743) | -0.63 (0.548) | -1.29 (0.736) | -0.84 (0.875)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 4, 8, 12, and 16
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. The LOCF method was used to impute missing post-Baseline FPG values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 4, Week 8, Week 12, and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Number analyzed (Participants) | 52 | 51 | 54 | 53
Millimoles per liter (mmol/L)
  Week 4 | 0.30 (1.190) | -1.54 (1.378) | -2.27 (1.465) | -1.32 (1.271)
  Week 8 | 0.41 (1.451) | -1.54 (1.585) | -2.27 (1.652) | -1.19 (1.458)
  Week 12 | 0.38 (1.612) | -1.25 (1.511) | -1.92 (1.388) | -1.06 (1.555)
  Week 16 | 0.50 (2.448) | -0.77 (1.583) | -1.92 (1.667) | -0.78 (1.821)

4. Secondary Outcome: Change From Baseline in Body Weight at Week 4, 8, 12, and 16
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The LOCF method was used to impute missing post-Baseline weight values.
Time Frame: Baseline; Week 4, Week 8, Week 12, and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Number analyzed (Participants) | 50 | 52 | 54 | 53
Kilograms
  Week 4 | -0.16 (0.956) | -0.36 (0.752) | -0.25 (1.268) | -0.02 (1.120)
  Week 8 | -0.29 (1.289) | -0.06 (0.926) | -0.46 (1.671) | -0.25 (1.684)
  Week 12 | -0.43 (1.409) | 0.09 (1.277) | -0.20 (1.906) | -0.22 (1.459)
  Week 16 | -0.65 (1.715) | 0.43 (1.468) | -0.20 (1.977) | -0.08 (1.740)

5. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5% and <7% at Weeks 4, 8, 12, and 16
Description: The number of participants who achieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5% and <7%) were assessed.
Time Frame: Week 4, Week 8, Week 12, and Week 16
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Number analyzed (Participants) | 50 | 52 | 54 | 53
Participants
  HbA1c <6.5%, Week 4 | 0 | 1 | 2 | 1
  HbA1c <6.5%, Week 8 | 0 | 5 | 15 | 5
  HbA1c <6.5%, Week 12 | 0 | 6 | 19 | 8
  HbA1c <6.5%, Week 16 | 0 | 5 | 18 | 8
  HbA1c <7%, Week 4 | 2 | 7 | 19 | 9
  HbA1c <7%, Week 8 | 4 | 12 | 27 | 18
  HbA1c <7%, Week 12 | 3 | 12 | 32 | 19
  HbA1c <7%, Week 16 | 3 | 9 | 34 | 21

6. Secondary Outcome: Mean Clearance of Albiglutide
Description: Clearance is defined as the volume of plasma cleared of albiglutide per unit time. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 1, 4, 5, 8, 12, and 13) and on the day of the clinic visit at Weeks 16, 20, and 24. At Weeks 0, 1, 4, 8, and 12, pharmacokinetic (PK) samples were collected immediately prior to dosing if a dose was scheduled for that week. At Weeks 16, 20, and 24, PK samples were collected at any time during the visit. The Week 5 post-dose PK sampling was performed any time between Weeks 4 and 6, within 2 to 5 days after administration of a dose; Week 13 post-dose PK sampling was performed any time between Weeks 12 and 14, within 2 to 5 days after administration of a dose of study medication. Modeled population PK data are presented; data were analyzed using a non-linear mixed effect modeling approach. A one-compartment PK model with first-order absorption and elimination processes was selected to describe GSK716155 PK.
Time Frame: Weeks 0, 1, 4, 5, 8, 12, 13, 16, 20, and 24
Population: PK Analysis Population: all participants for whom a PK sample was obtained and analyzed
Measure: Mean (95% Confidence Interval); unit: milliliters per hour
Groups:
- Albiglutide 15/30 mg Weekly or 30 mg Every Other Week: Participants received albiglutide 15 mg weekly, 30 mg weekly, or 30 mg or matching placebo administered via subcutaneous injection on alternating weeks via a fully disposable pen injector system for 16 weeks. The preferred post-rescue add-on treatment was insulin. Other medications may have been added at the investigator's discretion.
Arm/Group | Albiglutide 15/30 mg Weekly or 30 mg Every Other Week
Number analyzed (Participants) | 159
milliliters per hour | 47.8 [45.7 to 49.9]

7. Secondary Outcome: Mean Volume of Distribution of Albiglutide
Description: Volume of distribution is defined as the apparent volume in which albiglutide is distributed. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 1, 4, 5, 8, 12, and 13) and on the day of the clinic visit at Weeks 16, 20, and 24. At Weeks 0, 1, 4, 8, and 12, PK samples were collected immediately prior to dosing if a dose was scheduled for that week. At Weeks 16, 20, and 24, PK samples were collected at any time during the visit. The Week 5 post-dose PK sampling was performed any time between Weeks 4 and 6, within 2 to 5 days after administration of a dose; Week 13 post-dose PK sampling was performed any time between Weeks 12 and 14, within 2 to 5 days after administration of a dose of study medication. Modeled population PK data are presented; data were analyzed using a non-linear mixed effect modeling approach. A one-compartment PK model with first-order absorption and elimination processes was selected to describe GSK716155 PK.
Time Frame: Weeks 0, 1, 4, 5, 8, 12, 13, 16, 20, and 24
Population: PK Analysis Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Albiglutide 15/30 mg Weekly or 30 mg Every Other Week
Number analyzed (Participants) | 159
Liters | 9.34 [8.71 to 10.0]

8. Secondary Outcome: Mean Absorption Rate of Albiglutide
Description: Absorption rate is defined as the rate at which albiglutide enters the blood circulation. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 1, 4, 5, 8, 12, and 13) and on the day of the clinic visit at Weeks 16, 20, and 24. At Weeks 0, 1, 4, 8, and 12, PK samples were collected immediately prior to dosing if a dose was scheduled for that week. At Weeks 16, 20, and 24, PK samples were collected at any time during the visit. The Week 5 post-dose PK sampling was performed any time between Weeks 4 and 6, within 2 to 5 days after administration of a dose; Week 13 post-dose PK sampling was performed any time between Weeks 12 and 14, within 2 to 5 days after administration of a dose of study medication. Modeled population PK data are presented; data were analyzed using a non-linear mixed effect modeling approach. A one-compartment PK model with first-order absorption and elimination processes was selected to describe GSK716155 PK.
Time Frame: Weeks 0, 1, 4, 5, 8, 12, 13, 16, 20, and 24
Population: PK Analysis Population (Pop)
Measure: Mean (95% Confidence Interval); unit: hour^-1
Arm/Group | Albiglutide 15/30 mg Weekly or 30 mg Every Other Week
Number analyzed (Participants) | 159
hour^-1 | 0.0154 [0.0134 to 0.0183]

9. Secondary Outcome: Mean Half-maximal Effective Concentration (EC50) of Albiglutide for HbA1c and FPG
Description: EC50 is defined as the concentration of albiglutide that give a half-maximal HbA1c and FPG response. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 1, 4, 5, 8, 12, and 13) and on the day of the clinic visit at Weeks 16, 20, and 24. At Weeks 0, 1, 4, 8, and 12, PK samples were collected immediately prior to dosing if a dose was scheduled for that week. At Weeks 16, 20, and 24, PK samples were collected at any time during the visit. The Week 5 post-dose PK sampling was performed any time between Weeks 4 and 6, within 2 to 5 days after administration of a dose; Week 13 post-dose PK sampling was performed any time between Weeks 12 and 14, within 2 to 5 days after administration of a dose of study medication. EC50 estimates used PK data as well as HbA1c and FPG efficacy data. EC50 was estimated from an inhibitory Emax (maximal possible effect of albiglutide) model.
Time Frame: Weeks 0, 1, 4, 5, 8, 12, 13, 16, 20, and 24
Population: PK/PD Analysis Pop: all participants in the PK Analysis Pop with sufficient dosing history for inclusion in the PK/PD analysis. Modeled population PK data (analyzed using a non-linear mixed effect modeling approach) are presented. A one-compartment PK model with first-order absorption/elimination processes was selected to describe GSK716155 PK.
Measure: Mean (95% Confidence Interval); unit: nanograms per milliliter
Arm/Group | Albiglutide 15/30 mg Weekly or 30 mg Every Other Week
Number analyzed (Participants) | 157
nanograms per milliliter
  HbA1c | 3360 [2440 to 5260]
  FPG | 3850 [1420 to 6330]

ADVERSE EVENTS:
Time Frame: On-therapy serious adverse events (SAEs)/non-serious AEs, with a start date on/after the first day of study medication (SM) and within 56 days after the end of SM, were collected from the start of SM until Follow-up/Early Withdrawal (up to Study Day 168).
Description: On-therapy SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all enrolled participants who received at least one dose of study treatment. Participants were analyzed according to treatment received.
Arm/Group | Placebo | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 30 mg Every Other Week
Serious Adverse Events (participants affected / at risk) | 2/53 | 1/52 | 2/54 | 2/53
Other Adverse Events (participants affected / at risk) | 21/53 | 27/52 | 20/54 | 23/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Albiglutide 15 mg Weekly (N=52) | Albiglutide 30 mg Weekly (N=54) | Albiglutide 30 mg Every Other Week (N=53)
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Albiglutide 15 mg Weekly (N=52) | Albiglutide 30 mg Weekly (N=54) | Albiglutide 30 mg Every Other Week (N=53)
Nasopharyngitis (Infections and infestations) | 8 | 16 | 9 | 10
Cystitis (Infections and infestations) | 2 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 3 | 5
Constipation (Gastrointestinal disorders) | 1 | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Injection site reaction (General disorders) | 2 | 2 | 3 | 3
Injection site erythema (General disorders) | 0 | 2 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 3 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.